CLINICAL TRIAL: NCT06885671
Title: Phase II Single vs Hypofractionated Irradiation For Timely Access to Partial Breast Radiotherapy: SHIFT-PB
Brief Title: Single vs Hypofractionated Irradiation For Timely Access to Partial Breast Radiotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHIFT-PB
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)

STUDY DESIGN:
Intervention Model Description: This is a phase II randomized controlled trial, with the primary objective of testing feasibility of accruing 60 participants with early stage, node negative, breast cancer at 4 of the 6 BC Cancer centres and randomizing them to single vs. multiple fraction partial breast irradiation (PBI). Participants will be randomized 1:1 to 13Gy in 1 fraction vs 26 Gy in 5 fractions.
Who Masked: Outcomes Assessor
Masking Description: This will is an open-label randomized controlled study design, however, outcome assessors and data analysts will be blinded to the identity of each treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple Fraction PBI (Arm 1) (Active Comparator): For participants randomized to Arm 1, PBI will be delivered with a dose of 26 Gy in 5 daily fractions.
  Interventions: Radiation: Multiple Fraction PBI
- Single Fraction PBI (Arm 2) (Experimental): For participants randomized to Arm 2, PBI will be delivered in a single fraction with a dose of 13 Gy.
  Interventions: Radiation: Single Fraction PBI

INTERVENTIONS:
Radiation: Multiple Fraction PBI — Participants randomized to Arm 1 will receive PBI with a dose of 26 Gy in 5 daily fractions.
  Arms: Multiple Fraction PBI (Arm 1)
Radiation: Single Fraction PBI — Participants randomized to Arm 2 will receive PBI in a single fraction with a dose of 13 Gy.
  Arms: Single Fraction PBI (Arm 2)

SUMMARY:
Partial Breast Irradiation (PBI) is a targeted radiation approach commonly administered post-lumpectomy, specifically targeting the tumour bed. This targeted therapy reduces the exposure to other nearby tissues such as lungs, heart, and chest wall. However, traditional PBI treatment involves lengthy multiple fraction courses which presents a burden to patients from rural and remote communities, who must travel long distances to receive high quality cancer care. The purpose of this study is to compare single fraction (SF) PBI vs. multiple fraction (MF) PBI.

DETAILED DESCRIPTION:
Radiation can be delivered in multiple fractions, or doses, and can take up to several weeks or months of treatment depending on the type of cancer. Radiation can also be offered in a single fraction. Both techniques have evidence for use in clinical care. Multiple fraction is offered to reduce the amount of radiation given at a single time that could reduce late toxicities. However, single fraction radiotherapy is more cost-effective and saves patient time. With this trial, we will compare single fraction vs. multiple fraction PBI in regards to their impact on quality of life, rates of provider and participant reported toxicities, and local control.

ELIGIBILITY:
Inclusion Criteria:

* Female participants age 40 or older
* Able to provide informed consent
* pTis-2 pN0 cM0 breast cancer, with tumor size <3 cm as per provincial guidelines
* Able to complete electronic or paper entry of participant reported outcomes independently or with assistance from caregiver/family/friend/research staff
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* A history and physical examination, including ECOG performance status, performed within 8 weeks prior to enrollment.
* Participant is judged able to:

  * Maintain a stable position during therapy
  * Tolerate immobilization device(s) that may be required to deliver PBI safely
* Negative pregnancy test for People of Child-Bearing Potential (POCBP) within 4 weeks of RT start date

Exclusion Criteria:

* History of non-breast malignancies except adequately treated non-melanoma skin cancers, in situ cancers treated by local excision or other cancers curatively treated with no evidence of disease for ≥ 5 years.
* Uncontrolled concurrent malignant cancer
* Seroma not visible
* Ipsilateral implanted cardiac device
* Prior radiotherapy requiring summation for planning.
* Inability to meet mandatory planning constraints.
* Requirement for a radiation boost (as determined by the treating investigator)
* Positive surgical margins
* Surgical cavities lacking clear delineation (surgical clips are not required but may assist in target delineation)
* Known germline BRCA1/2 mutation.
* Serious medical comorbidities precluding radiotherapy (e.g., connective tissue disorders such as lupus or scleroderma)
* Pregnant or breastfeeding

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants must be biologically female.
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants accrued | 2 years
  Number of participants who sign consent to be randomized to 1 vs 5 fractions of radiotherapy for PBI over a 2 year period

SECONDARY OUTCOMES:
Time from CT simulation to plan approval | Baseline
  Measured as the time from the day of CT simulation to the date of plan approval.
2-Year Local Control Rates | 6 weeks, 6 months, 12, months, 18 months, and 24 months post-treatment
  Absence of ipsilateral in-breast recurrence, defined as histologic evidence of invasive or in situ breast cancer in the ipsilateral breast 2 years post-treatment
Quality of life assessed using the POSI-Breast questionnaire | Baseline, 6 weeks, 6 months, 12 months, 18 months, and 24 months post treatment
  Prospective Outcomes and Support Initiative (POSI) for Breast Data will be used to measure and compare the quality of life of participants in both arms.
Rates of provider-rated toxicities: Occurrences of adverse events as measured by CTCAE | Baseline, 6 weeks, 6 months, 12 months, 18 months, and 24 months post treatment
  Participant-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Data will be used to measure and compare participant-reported toxicities in both arms.
Participant-reported toxicities | Baseline, 6 weeks, 6 months, 12, months, 18 months, and 24 months post-treatment
  Occurrences of adverse events as measured by PRO-CTCAE
Overall Survival (OS) | Approximately at the end of year 2 (study completion)
  Time from randomization to death from any cause, or last follow-up, whichever occurs first.
Progression-Free Survival (PFS) | 6 weeks, 6 months, 12 months, 18 months, and approximately at the end of 24 months
  Time from randomization to disease progression at any site, death, or last follow-up, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olson, MD, MSc, FRCPC, Principal Investigator — BC Cancer - Prince George

REFERENCES:
- [Derived] Olson R, Cua M, Matthews Q, Laing J, Narinesingh D, Nichol A, Berrang T, Koulis T, Karan T, Chng N. Phase II single vs hypofractionated irradiation for timely access to partial breast radiotherapy (SHIFT-PB). BMC Cancer. 2025 Aug 8;25(1):1285. doi: 10.1186/s12885-025-14720-w. PMID 40781619